CLINICAL TRIAL: NCT02357498
Title: Prospective Multicenter Cohort Study Comparing Extent of Tumor Resection Between Microscopic Transsphenoidal Surgery and Fully Endoscopic Transsphenoidal Surgery for Nonfunctioning Pituitary Adenomas
Brief Title: Transsphenoidal Extent of Resection Study
Acronym: TRANSSPHER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Saint John's Cancer Institute (Other); Swedish Medical Center (Other); Northwestern University (Other); Ohio State University (Other); Washington University School of Medicine (Other); University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, Pam Dewey, Clinical Research Operations Manager, St. Joseph's Hospital and Medical Center, Phoenix
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14BN151
Record Dates: First submitted 2015-01-26; First posted 2015-02-06 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Pituitary Adenoma
Keywords: pituitary; adenoma; transsphenoidal surgery
MeSH Terms: conditions — Pituitary Neoplasms; Pituitary Diseases; Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- microscopic (Active Comparator): Microscopic transsphenoidal surgery, including endoscopic-assisted approach (350 subjects)
  Interventions: Procedure: transsphenoidal surgery
- endoscopic (Active Comparator): Fully endoscopic transsphenoidal surgery (350 subjects)
  Interventions: Procedure: transsphenoidal surgery

INTERVENTIONS:
Procedure: transsphenoidal surgery

SUMMARY:
The purpose of this research study is to compare the extent of resection (EOR) in patients with nonfunctioning pituitary adenomas undergoing transsphenoidal surgery using a microsurgical technique to those patients who have undergone surgery with a fully endoscopic technique. Another goal is to compare surgical complications, endocrine outcomes, visual outcomes, length of surgery, length of hospital stay, and readmission rates between the two transsphenoidal surgery techniques. This is an observational data collection study with no experimental procedures or experimental medicines. Endonasal transsphenoidal removal of a pituitary tumor is a unique procedure and there is little information comparing the two surgical techniques.

DETAILED DESCRIPTION:
The treatment of choice for most patients with symptomatic nonfunctioning pituitary adenomas is transsphenoidal surgery to improve vision by decompression of the optic chiasm, to prevent the development of endocrine dysfunction, and to treat neurological symptoms such as headache or cranial neuropathies caused by the tumor. The most widely accepted surgical technique is microscopic transsphenoidal surgery, in which an operating microscope is used by the surgeon to provide surgical visualization and a nasal speculum is used to maintain the operative corridor. [1-4] Recently, fully endoscopic transsphenoidal surgery, in which surgical visualization is achieved using an endoscope, has been adopted by many pituitary surgeons because the technique offers superior panoramic and angled visualization of the surgical target and may permit greater tumor resection. [5-10] There is a vigorous debate in the neurosurgical community about the relative merits of the microscopic and endoscopic techniques. Proponents of the endoscopic technique argue that the superior visualization permits more aggressive tumor resection and better preservation of the normal pituitary gland. Proponents of the microscopic technique argue that it permits shorter operative times, results in similar surgical outcomes, and has a lower complication rate.

Despite the adoption of fully endoscopic surgery by many surgeons, no prospective studies have compared the extent of tumor resection (EOR) between microscopic and endoscopic approaches. Numerous retrospective studies have established the efficacy of each approach, but only a few studies present comparative data.[11-13] Recently, McLaughlin et al. noted that the addition of endoscopy to microscopic pituitary surgery enhances tumor removal, particularly in patients with tumors greater than 20 mm in diameter. [14] This study raises the intriguing possibility that certain subgroups of patients (e.g. patients with larger tumors) may benefit from endoscopic surgery. In patients with smaller tumors with no cavernous sinus invasion, others have shown that the techniques achieve similar EOR. [15] That endoscopy may permit more complete tumor resections is a testable hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected nonfunctioning pituitary macroadenomas (≥ 1 cm) with planned transsphenoidal surgery
* Adults (age 18-80 years)
* Medically stable for surgery
* Reasonable expectation that patient will complete study and be available for follow-up assessments

Exclusion Criteria:

* Prisoners
* Pregnant women
* Patients with suspected functioning pituitary adenoma
* Unable to obtain MRI of the pituitary (e.g., pacemaker, anaphylaxis to gadolinium, low GFR)
* Pituitary apoplexy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
percentage of patients who have complete tumor removal (gross total resection) based on MRI . | 3 months post surgery
  Postop MRI read by neuroradiologist

SECONDARY OUTCOMES:
volume of residual tumor | 3 months after date of surgery
  volume, analyzed as a continuous variable; will be determined by manual segmentation using Dominator (www.dominator.com) software under the supervision of a board-certified neuroradiologist
percentage of tumor removed | 3 months post surgery
  Postop MRI tumor bed read by neuroradilogisy
postoperative cerebral-spinal fluid (CSF) leak | 6 months (continuous) from surgery
  leakage from nose is a known complication, however, patients who have undergone a second surgery or had a lumbar drain placed to repair the problem will be documented
postoperative meningitis | 6 months (continuous) from surgery
  Determined by symptoms of headache, fever, neck stiffness, nausea and vomiting, and occasionally an altered level of consciousness. CSF culture may be positive for infection and may show elevated glucose and/or protein. CSF may be negative in aseptic meningitis.
hypopituitarism | 6 months post surgery
  (morning cortisol <4.0ug/dL)(adrenocorticotropic hormone ACTH <6.0pg/mL)(follicular stimulating hormone FSH - mIU/mL. Female: follicular: <3.5; midcycle <4.7; luteal <1.7; postmenopausal <25.8. male <1.7)(luteinizing hormone LH - mIU/mL. Female: follicular <2.4; midcycle <14.0; luteal <1.0; postmenopausal <7.7)(estradiol - pg/mL. female: follicular <13; ovulation <86; luteal <44; postmenopausal <56)(insulin-like growth factor 1 IGF1: 101ng/mL)(testosterone total - ng/dL. Female <6.0; male <270.0)(prolactin ,3.3ng/mL)(thyroid stimulating hormone TSH <.45mU/L)(Thyroxine T4 Free <0.8ng/dL
diabetes insipidus (DI) | 6 months post surgery
  to be evaluated by pituitary endocrinologist; serum sodium value is > or equal to 147meq/dl OR if the patient received treatment for DI
visual outcomes | 3 months post surgery
  visual field deficits in this exam will be compared to pre-operative results. Confrontation visual field exam (Donder's test): The examiner will ask the patient to cover one eye and stare at the examiner. The examiner will then move his hand out of the patient's visual field and bring it back in. The examiner will use a slowly wagging finger or a hat pin for this. The patient signals the examiner when his hand comes back into view. Second option is a formal visual field exam (perimetry) performed by a neuro-ophthalmologist.
hypothyroidism | 6 months post surgery
  (thyroid stimulating hormone TSH <.45mU/L)(thyroxine T4Free <0.8ng/dL)
hypogonadism | 6 months post surgery
  (Testosterone (Total) - ng/dL. Female: < 6.0; Male: < 270.0) (Follicular Stimulating Hormone (FSH) - mIU/mL. Female - Follicular: < 3.5; Midcycle: <4.7; Luteal: < 1.7; Postmenopausal: < 25.8. Male - < 1.5)(Luteinizing Hormone LH - mIU/mL. Female: Follicular: < 2.4; Midcycle: <14.0; Luteal: < 1.0; Postmenopausal: < 7.7. Male: < 1.7)(Estradiol - pg/mL. Female: Follicular: < 13; Ovulation: < 86; Luteal: < 44; Postmenopausal: < 56. Male: < 15)
growth hormone deficiency | 6 months post surgery
  (insulin tolerance test: growth hormone <3μg/l)(IGF1 <77)(symptoms may include thin and dry skin, low energy, decreased strength and exercise tolerance, decreased muscle mass, weight gain especially around the waist, feelings of anxiety, depression, or sadness causing a change in social behavior
adrenal insufficiency | 6 months post surgery
  (morning serum cortisol <4.0ug/dL)(ACTH <6.0pg/mL)(sodium <135mEq/L)(abnormal ACTH [cosyntropin] stimulation test)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Little, MD, Principal Investigator — Saint Joseph's Hospital and Medical Center/Barrow Neurological Institute
Locations (7):
- United States (7):
  - Barrow Neurological Institute/St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Northwestern University, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Ohio State University Medical Center, Columbus, Ohio
  - Swedish Neuroscience Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson CB, Rand RW, Grollmus JM, Heuser G, Levin S, Goldfield E, Schneider V, Linfoot J, Hosobuchi Y. Surgical experience with a microscopic transsphenoidal approach to pituitary tumors and non-neoplastic parasellar conditions. Calif Med. 1972 Nov;117(5):1-9. PMID 4638402
- [Background] Hardy J. Transsphenoidal hypophysectomy. J Neurosurg. 1971 Apr;34(4):582-94. doi: 10.3171/jns.1971.34.4.0582. No abstract available. PMID 5554367
- [Background] Fatemi N, Dusick JR, de Paiva Neto MA, Kelly DF. The endonasal microscopic approach for pituitary adenomas and other parasellar tumors: a 10-year experience. Neurosurgery. 2008 Oct;63(4 Suppl 2):244-56; discussion 256. doi: 10.1227/01.NEU.0000327025.03975.BA. PMID 18981830
- [Background] Patel SK, Husain Q, Eloy JA, Couldwell WT, Liu JK. Norman Dott, Gerard Guiot, and Jules Hardy: key players in the resurrection and preservation of transsphenoidal surgery. Neurosurg Focus. 2012 Aug;33(2):E6. doi: 10.3171/2012.6.FOCUS12125. PMID 22853837
- [Background] Dehdashti AR, Ganna A, Karabatsou K, Gentili F. Pure endoscopic endonasal approach for pituitary adenomas: early surgical results in 200 patients and comparison with previous microsurgical series. Neurosurgery. 2008 May;62(5):1006-15; discussion 1015-7. doi: 10.1227/01.neu.0000325862.83961.12. PMID 18580798
- [Background] Gondim JA, Schops M, de Almeida JP, de Albuquerque LA, Gomes E, Ferraz T, Barroso FA. Endoscopic endonasal transsphenoidal surgery: surgical results of 228 pituitary adenomas treated in a pituitary center. Pituitary. 2010;13(1):68-77. doi: 10.1007/s11102-009-0195-x. Epub 2009 Aug 21. PMID 19697135
- [Background] Cavallo LM, Prevedello DM, Solari D, Gardner PA, Esposito F, Snyderman CH, Carrau RL, Kassam AB, Cappabianca P. Extended endoscopic endonasal transsphenoidal approach for residual or recurrent craniopharyngiomas. J Neurosurg. 2009 Sep;111(3):578-89. doi: 10.3171/2009.2.JNS081026. PMID 19326977
- [Background] Cavallo LM, Prevedello D, Esposito F, Laws ER Jr, Dusick JR, Messina A, Jane JA Jr, Kelly DF, Cappabianca P. The role of the endoscope in the transsphenoidal management of cystic lesions of the sellar region. Neurosurg Rev. 2008 Jan;31(1):55-64; discussion 64. doi: 10.1007/s10143-007-0098-0. Epub 2007 Oct 6. PMID 17922153
- [Background] Jho HD, Alfieri A. Endoscopic endonasal pituitary surgery: evolution of surgical technique and equipment in 150 operations. Minim Invasive Neurosurg. 2001 Mar;44(1):1-12. doi: 10.1055/s-2001-13590. PMID 11409304
- [Background] Jho HD, Carrau RL. Endoscopic endonasal transsphenoidal surgery: experience with 50 patients. J Neurosurg. 1997 Jul;87(1):44-51. doi: 10.3171/jns.1997.87.1.0044. PMID 9202264
- [Background] Ammirati M, Wei L, Ciric I. Short-term outcome of endoscopic versus microscopic pituitary adenoma surgery: a systematic review and meta-analysis. J Neurol Neurosurg Psychiatry. 2013 Aug;84(8):843-9. doi: 10.1136/jnnp-2012-303194. Epub 2012 Dec 15. PMID 23243265
- [Background] Starke RM, Raper DM, Payne SC, Vance ML, Oldfield EH, Jane JA Jr. Endoscopic vs microsurgical transsphenoidal surgery for acromegaly: outcomes in a concurrent series of patients using modern criteria for remission. J Clin Endocrinol Metab. 2013 Aug;98(8):3190-8. doi: 10.1210/jc.2013-1036. Epub 2013 Jun 4. PMID 23737543
- [Background] McLaughlin N, Eisenberg AA, Cohan P, Chaloner CB, Kelly DF. Value of endoscopy for maximizing tumor removal in endonasal transsphenoidal pituitary adenoma surgery. J Neurosurg. 2013 Mar;118(3):613-20. doi: 10.3171/2012.11.JNS112020. Epub 2012 Dec 14. PMID 23240699
- [Background] Dallapiazza R, Bond AE, Grober Y, Louis RG, Payne SC, Oldfield EH, Jane JA Jr. Retrospective analysis of a concurrent series of microscopic versus endoscopic transsphenoidal surgeries for Knosp Grades 0-2 nonfunctioning pituitary macroadenomas at a single institution. J Neurosurg. 2014 Sep;121(3):511-7. doi: 10.3171/2014.6.JNS131321. Epub 2014 Jul 4. PMID 24995783
- [Background] Little AS, Kelly D, Milligan J, Griffiths C, Rosseau G, Prevedello DM, Carrau R, Jahnke H, Chaloner C, O'Leary J, Chapple K, Nakaji P, White WL. Prospective validation of a patient-reported nasal quality-of-life tool for endonasal skull base surgery: The Anterior Skull Base Nasal Inventory-12. J Neurosurg. 2013 Oct;119(4):1068-74. doi: 10.3171/2013.3.JNS122032. Epub 2013 May 10. PMID 23662829
- [Background] Gao Y, Zhong C, Wang Y, Xu S, Guo Y, Dai C, Zheng Y, Wang Y, Luo Q, Jiang J. Endoscopic versus microscopic transsphenoidal pituitary adenoma surgery: a meta-analysis. World J Surg Oncol. 2014 Apr 11;12:94. doi: 10.1186/1477-7819-12-94. PMID 24721812
- [Background] Goudakos JK, Markou KD, Georgalas C. Endoscopic versus microscopic trans-sphenoidal pituitary surgery: a systematic review and meta-analysis. Clin Otolaryngol. 2011 Jun;36(3):212-20. doi: 10.1111/j.1749-4486.2011.02331.x. PMID 21752205
- [Background] Rudmik L, Starreveld YP, Vandergrift WA, Banglawala SM, Soler ZM. Cost-effectiveness of the endoscopic versus microscopic approach for pituitary adenoma resection. Laryngoscope. 2015 Jan;125(1):16-24. doi: 10.1002/lary.24780. Epub 2014 Jun 17. PMID 24938934
- [Background] Tabaee A, Anand VK, Barron Y, Hiltzik DH, Brown SM, Kacker A, Mazumdar M, Schwartz TH. Endoscopic pituitary surgery: a systematic review and meta-analysis. J Neurosurg. 2009 Sep;111(3):545-54. doi: 10.3171/2007.12.17635. PMID 19199461
- [Background] Zhu M, Yang J, Wang Y, Cao W, Zhu Y, Qiu L, Tao Y, Xu Y, Xu H. [Endoscopic transsphenoidal surgery versus microsurgery for the resection of pituitary adenomas: a systematic review]. Zhonghua Er Bi Yan Hou Tou Jing Wai Ke Za Zhi. 2014 Mar;49(3):236-9. Chinese. PMID 24820497
- [Background] Komotar RJ, Starke RM, Raper DM, Anand VK, Schwartz TH. Endoscopic endonasal compared with microscopic transsphenoidal and open transcranial resection of craniopharyngiomas. World Neurosurg. 2012 Feb;77(2):329-41. doi: 10.1016/j.wneu.2011.07.011. Epub 2011 Nov 1. PMID 22501020
- [Result] Little AS, Gardner PA, Fernandez-Miranda JC, Chicoine MR, Barkhoudarian G, Prevedello DM, Yuen KCJ, Kelly DF; TRANSSPHER Study Group. Pituitary gland recovery following fully endoscopic transsphenoidal surgery for nonfunctioning pituitary adenoma: results of a prospective multicenter study. J Neurosurg. 2019 Nov 15;133(6):1732-1738. doi: 10.3171/2019.8.JNS191012. Print 2020 Dec 1. PMID 31731279
- [Result] Little AS, Chicoine MR, Kelly DF, Sarris CE, Mooney MA, White WL, Gardner PA, Fernandez-Miranda JC, Barkhoudarian G, Chandler JP, Prevedello DM, Liebelt BD, Sfondouris J, Mayberg MR; TRANSSPHER Study Group. Evaluation of Surgical Resection Goal and Its Relationship to Extent of Resection and Patient Outcomes in a Multicenter Prospective Study of Patients With Surgically Treated, Nonfunctioning Pituitary Adenomas: A Case Series. Oper Neurosurg. 2020 Jan 1;18(1):26-33. doi: 10.1093/ons/opz085. PMID 31079156
- [Result] Little AS, Kelly DF, White WL, Gardner PA, Fernandez-Miranda JC, Chicoine MR, Barkhoudarian G, Chandler JP, Prevedello DM, Liebelt BD, Sfondouris J, Mayberg MR; TRANSSPHER Study Group. Results of a prospective multicenter controlled study comparing surgical outcomes of microscopic versus fully endoscopic transsphenoidal surgery for nonfunctioning pituitary adenomas: the Transsphenoidal Extent of Resection (TRANSSPHER) Study. J Neurosurg. 2019 Mar 22;132(4):1043-1053. doi: 10.3171/2018.11.JNS181238. Print 2020 Apr 1. PMID 30901746
- [Result] Mooney MA, Sarris CE, Zhou JJ, Barkhoudarian G, Chicoine MR, Fernandez-Miranda JC, Gardner PA, Hardesty DA, Jahnke H, Kelly DF, Liebelt BD, Mayberg MR, Prevedello DM, Sfondouris J, Sheehy JP, Chandler JP, Yuen KCJ, White WL, Little AS; TRANSSPHER Study Group. Proposal and Validation of a Simple Grading Scale (TRANSSPHER Grade) for Predicting Gross Total Resection of Nonfunctioning Pituitary Macroadenomas After Transsphenoidal Surgery. Oper Neurosurg. 2019 Nov 1;17(5):460-469. doi: 10.1093/ons/opy401. PMID 30649445
- [Result] Mooney MA, Herro AM, Fintelmann RE, Mayberg MR, Barkhoudarian G, Gardner PA, Prevedello DM, Chicoine MR, Kelly DF, Chandler JP, Jahnke H, White WL, Little AS. Visual Field Outcome Reporting in Neurosurgery: Lessons Learned from a Prospective, Multicenter Study of Transsphenoidal Pituitary Surgery. World Neurosurg. 2018 Dec;120:e326-e332. doi: 10.1016/j.wneu.2018.08.069. Epub 2018 Aug 23. PMID 30144606